CLINICAL TRIAL: NCT00039130
Title: Phase II Study Of Rituximab And Short Duration, High Intensity Chemotherapy With G-CSF Support In Previously Untreated Patients With Burkitt Lymphoma/Leukemia
Brief Title: Rituximab, Chemotherapy, and Filgrastim in Treating Patients With Burkitt's Lymphoma or Burkitt's Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-10002; U10CA031946 (NIH); CALGB-10002; CDR0000069354 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Rituximab; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Prednisone; Vincristine; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab with High Intensity Chemotherapy (Experimental): Cycle1: Cyclophosphamide 100 mg/m^2/day (d) IV (d 1-5), Prednisone 60 mg/m^2/d oral (d 1-7), Allopurinal 300 mg/d oral (d 1-14) Cycle 2, 4 & 6 (21 day): Ifosfamide 800 mg/m^2/d (d 1-5), Dexamethasone 10 mg/m^2/d (d1-5), Methotrexate 150 mg/m^2 load, then 1.35 g/m^2 over 23.5 h (d 1), Leucovorin 25 mg/m^2 36 h after methotrexate (d 2) then 10 mg/m^2 every 6 h, Vincristine 2 mg push (d 1), Cytarabine 1000 mg/m^2/d over 2 h (d 4-5), Etoposide 80 mg/m^2.d over 1 h (d 4-5), Filgrastim 5 mg/kg/d (d 7-21 as needed), Rituximab 50 mg/m^2 d 8 cycle 2 only, 375 mg/m^2/d (d 10, 12 cycle 2, d 8 cycle 4 & 6) Cycle 3, 5 & 7 (21 day): Cyclophosphamide 200 mg/m^2/day (d) IV (d 1-5), Dexamethasone 10 mg/m^2/d (d1-5), Methotrexate 150 mg/m^2 load, then 1.35 g/m^2 over 23.5 h (d 1), Leucovorin 50 mg/m^2 36 h after methotrexate (d 2) then 10 mg/m^2 every 6 h, Vincristine 2 mg push (d 1), Doxorubicin 25 mg/m^2/d (d 4-5), Filgrastim 5 mg/kg/d (d 7-21 as needed), Rituximab 375 mg/m^2/d (d 8)
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Drug: Allopurinol

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg/day sub Q injection day 7 until ANC>5000/ul courses II-VII
Biological: rituximab — Day 8 course II 50 mg/sq m IV infusion: d 8 course IV & VI 375mg/sq m IV Day 10 course II: 325 mg/sq m IV infusion Day 12 course II: 375 mg/sq m IV infusion
Drug: cyclophosphamide — 200 mg/sq m/day IV infusion over 5-15 min days 1-5, courses I, III, V, VII
Drug: cytarabine — 1 g/sq m/day IV infusion Days 4 & 5, courses II, IV, VI
Drug: dexamethasone — 10mg/sq m PO or IV Days 1-5 courses II-VII
Drug: doxorubicin hydrochloride — 25 mg/sq m/day IV infusion Days 4 & 5 courses III,V, VII
Drug: etoposide — 80 mg/sq m/day IV infusion Days 4 & 5 courses II, IV, VI
Drug: ifosfamide — 800 mg/sq m/day IV infusion Days 1-5 courses II, IV, VI
Drug: leucovorin calcium — 25mg/sq m IV infusion over 15 min then 10 mg IV q 6 hrs until serum MTX <10nM, courses II-VII
Drug: methotrexate — 1.5 g/sq m IV infusion Day 1 courses II-VII
Drug: prednisone — 60 mg/sq m PO/day Days 1-7 course I
Drug: vincristine sulfate — 2 mg IV push Day 1 courses II-VII
Drug: Allopurinol — 300 mg/day PO Days 1-14, course I

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the numbers of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Combining chemotherapy with rituximab and filgrastim may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab with chemotherapy and filgrastim in treating patients who have Burkitt's lymphoma or Burkitt's leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate in patients with previously untreated Burkitt's lymphoma or Burkitt's leukemia treated with rituximab and high-intensity chemotherapy with filgrastim (G-CSF) support.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the feasibility and toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (leukemia vs lymphoma).

* Course 1: Patients receive cyclophosphamide IV over 5-15 minutes daily on days 1-5 and oral prednisone on days 1-7. Allopurinol PO will be given on days 1-14.
* Courses 2, 4, and 6: Patients receive ifosfamide IV over 1 hour daily on days 1-5; vincristine IV over 10 minutes and methotrexate IV over 24 hours on day 1; leucovorin calcium IV over 15 minutes every 6 hours on day 2; cytarabine IV over 2 hours on days 4 and 5 and etoposide IV over 1 hour daily on days 4 and 5; oral dexamethasone daily on days 1-5; and methotrexate and cytarabine intrathecally (IT) on day 1. During course 2, patients receive rituximab IV over 1-4 hours on days 8, 10, and 12. During courses 4 and 6, patients receive rituximab IV over 1 hour on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 7 and continuing until blood counts recover.
* Courses 3, 5, and 7: Patients receive cyclophosphamide IV over 5-15 minutes daily on days 1-5; vincristine IV over 10 minutes and methotrexate IV over 24 hours on day 1; leucovorin calcium IV every 6 hours on day 2; doxorubicin IV daily on days 4 and 5; oral dexamethasone daily on days 1-5; methotrexate and cytarabine IT on day 1; and rituximab IV over 1 hour on day 8. Patients also receive G-CSF as in courses 2, 4, and 6. After course 3, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 100 patients (50 per stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically, cytogenetically, or immunophenotypically confirmed Burkitt's leukemia or Burkitt's or Burkitt-like lymphoma

  * L3 morphology surface IgG expression
  * Cytogenetic evidence for t(8;14), t(8;22), or t(2;8)
* Previously untreated disease except hydroxyurea for leukocytosis
* CNS involvement allowed
* Patients with Burkitt's leukemia or Burkitt's lymphoma with bone marrow involvement must also be enrolled on CALGB-8461
* Patients with Burkitt's leukemia must also be enrolled on CALGB-9665

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent interleukin-11

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except for non-disease-related conditions (e.g., insulin for diabetes)
* No concurrent steroids except for adrenal failure

Radiotherapy:

* No concurrent palliative radiotherapy except whole-brain irradiation for documented CNS disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2002-05; Primary Completion 2010-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Study Chair — Duke University Medical Center Bone Marrow Transplant
Locations (31):
- United States (31):
  - Naval Medical Center - San Diego, San Diego, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Rizzieri DA, Johnson JL, Byrd JC, Lozanski G, Blum KA, Powell BL, Shea TC, Nattam S, Hoke E, Cheson BD, Larson RA; Alliance for Clinical Trials In Oncology (ACTION). Improved efficacy using rituximab and brief duration, high intensity chemotherapy with filgrastim support for Burkitt or aggressive lymphomas: cancer and Leukemia Group B study 10 002. Br J Haematol. 2014 Apr;165(1):102-11. doi: 10.1111/bjh.12736. Epub 2014 Jan 15. PMID 24428673

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab With High Intensity Chemotherapy
Started | 105
Completed | 75
Not Completed | 30
Not completed — Adverse Event | 11
Not completed — Death | 9
Not completed — Withdrawal by Subject | 3
Not completed — Progression | 2
Not completed — Subsequent treatment | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab With High Intensity Chemotherapy
Number analyzed (Participants) | 105
Age, Continuous [Median (Full Range); unit: years] | 43 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 98
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Response is assessed by investigator according to Revised Response Criteria for Malignant Lymphoma. Complete response requires disappearance of all evidence of disease.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab With High Intensity Chemotherapy
Number analyzed (Participants) | 105
percentage of participants | 83 [74 to 90]

2. Secondary Outcome: 2 Year Event Free Survival
Description: Percentage of patients who were event free at 2 years. The 2-year event free rate was estimated using the Kaplan Meier method. An event is defined as death, progression or treatment failure.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab With High Intensity Chemotherapy
Number analyzed (Participants) | 105
percentage of participants | 78 [69 to 85]

3. Secondary Outcome: 2 Year Overall Survival
Description: Percentage of participants who were alive at 2 years. The 2 year survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab With High Intensity Chemotherapy
Number analyzed (Participants) | 105
percentage of participants | 80 [71 to 86]

ADVERSE EVENTS:
Arm/Group | Rituximab With High Intensity Chemotherapy
Serious Adverse Events (participants affected / at risk) | 61/105
Other Adverse Events (participants affected / at risk) | 101/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab With High Intensity Chemotherapy (N=105)
Febrile neutropenia (Blood and lymphatic system disorders) | 31 (40)
Hemoglobin decreased (Blood and lymphatic system disorders) | 58 (81)
Lymphatic disorder (Blood and lymphatic system disorders) | 2 (2)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Transfusion: Platelets (Blood and lymphatic system disorders) | 3 (3)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 5 (6)
Arrhythmia (Cardiac disorders) | 4 (4)
Arrhythmia supraventricular (Cardiac disorders) | 4 (4)
Cardiac disorder (Cardiac disorders) | 3 (3)
Conduction disorder (Cardiac disorders) | 2 (2)
Edema (Cardiac disorders) | 20 (21)
Left ventricular failure (Cardiac disorders) | 4 (4)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 11 (13)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 12 (13)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (5)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhea (Gastrointestinal disorders) | 27 (30)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 28 (34)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3)
Melena/GI bleeding (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 45 (59)
Nausea (Gastrointestinal disorders) | 32 (41)
Oral pain (Gastrointestinal disorders) | 4 (4)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 5 (6)
Rectal pain (Gastrointestinal disorders) | 2 (4)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (25)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 10 (12)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 31 (37)
Fever (General disorders) | 11 (11)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 24 (27)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (4)
Infection (Infections and infestations) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 32 (36)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 19 (20)
Infectious colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound-infectious (Infections and infestations) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 7 (8)
Alanine aminotransferase increased (Investigations) | 28 (36)
Alkaline phosphatase (Investigations) | 17 (21)
Alkaline phosphatase increased (Investigations) | 3 (3)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 25 (32)
Blood bilirubin increased (Investigations) | 22 (23)
Cardiac troponin I increased (Investigations) | 2 (2)
Coagulopathy (Investigations) | 2 (2)
Creatinine increased (Investigations) | 26 (29)
INR increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 7 (8)
Leukocyte count decreased (Investigations) | 19 (26)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 13 (16)
Neutrophil count decreased (Investigations) | 55 (72)
Platelet count decreased (Investigations) | 56 (75)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 7 (7)
Acidosis (Metabolism and nutrition disorders) | 4 (4)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 16 (18)
Blood glucose increased (Metabolism and nutrition disorders) | 47 (63)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 4 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 23 (31)
Serum calcium decreased (Metabolism and nutrition disorders) | 32 (40)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 20 (25)
Serum magnesium increased (Metabolism and nutrition disorders) | 5 (5)
Serum phosphate decreased (Metabolism and nutrition disorders) | 12 (12)
Serum potassium decreased (Metabolism and nutrition disorders) | 40 (49)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 15 (20)
Serum sodium increased (Metabolism and nutrition disorders) | 7 (7)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7)
Encephalopathy (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 19 (22)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 6 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (13)
Seizure (Nervous system disorders) | 3 (3)
Speech disorder (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (8)
Confusion (Psychiatric disorders) | 8 (8)
Depression (Psychiatric disorders) | 9 (9)
Insomnia (Psychiatric disorders) | 3 (3)
Personality change (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (2)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (7)
Urethral fistula (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 5 (5)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 14 (15)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 8 (8)
Flushing (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 2 (2)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 10 (10)
Hypotension (Vascular disorders) | 14 (17)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab With High Intensity Chemotherapy (N=105)
Blood disorder (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 65 (130)
Hemoglobin decreased (Blood and lymphatic system disorders) | 100 (642)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Transfusion: Platelets (Blood and lymphatic system disorders) | 18 (41)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 18 (72)
Arrhythmia (Cardiac disorders) | 4 (4)
Arrhythmia supraventricular (Cardiac disorders) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac disorder (Cardiac disorders) | 10 (10)
Edema (Cardiac disorders) | 38 (80)
Left ventricular failure (Cardiac disorders) | 3 (5)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 11 (12)
Sinus tachycardia (Cardiac disorders) | 22 (35)
Ear disorder (Ear and labyrinth disorders) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 4 (4)
Diplopia (Eye disorders) | 2 (3)
Dry eye syndrome (Eye disorders) | 5 (6)
Eye disorder (Eye disorders) | 9 (12)
Flashing vision (Eye disorders) | 3 (3)
Photophobia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 10 (15)
Watering eyes (Eye disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 43 (78)
Anal fistula (Gastrointestinal disorders) | 3 (4)
Anal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 53 (111)
Diarrhea (Gastrointestinal disorders) | 63 (127)
Dry mouth (Gastrointestinal disorders) | 12 (14)
Dyspepsia (Gastrointestinal disorders) | 24 (39)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 6 (6)
Esophageal pain (Gastrointestinal disorders) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 59 (121)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 12 (14)
Hemorrhoids (Gastrointestinal disorders) | 2 (4)
Ileus (Gastrointestinal disorders) | 2 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 5 (6)
Mucositis oral (Gastrointestinal disorders) | 91 (325)
Nausea (Gastrointestinal disorders) | 89 (294)
Oral pain (Gastrointestinal disorders) | 6 (8)
Proctitis (Gastrointestinal disorders) | 2 (2)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 5 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 10 (16)
Vomiting (Gastrointestinal disorders) | 53 (121)
Chest pain (General disorders) | 7 (8)
Chills (General disorders) | 21 (28)
Edema limbs (General disorders) | 8 (12)
Fatigue (General disorders) | 79 (279)
Fever (General disorders) | 26 (39)
General symptom (General disorders) | 8 (9)
Ill-defined disorder (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 49 (113)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 4 (7)
Hypersensitivity (Immune system disorders) | 6 (8)
Immune system disorder (Immune system disorders) | 2 (4)
Abdominal infection (Infections and infestations) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 6 (9)
Infection (Infections and infestations) | 8 (12)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 65 (144)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 51 (101)
Mucosal infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound-infectious (Infections and infestations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 5 (5)
Operative injury to bladder and/or ureter (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 12 (17)
Alanine aminotransferase increased (Investigations) | 71 (236)
Alkaline phosphatase (Investigations) | 46 (92)
Alkaline phosphatase increased (Investigations) | 16 (29)
Amylase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 66 (175)
Blood bilirubin increased (Investigations) | 41 (89)
Coagulopathy (Investigations) | 4 (4)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 46 (139)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
Fibrinogen decreased (Investigations) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (6)
INR increased (Investigations) | 11 (20)
Laboratory test abnormal (Investigations) | 17 (34)
Leukocyte count decreased (Investigations) | 45 (169)
Lymphocyte count decreased (Investigations) | 36 (137)
Neutrophil count decreased (Investigations) | 98 (493)
Platelet count decreased (Investigations) | 98 (596)
Serum cholesterol increased (Investigations) | 2 (4)
Weight gain (Investigations) | 5 (5)
Weight loss (Investigations) | 21 (22)
Anorexia (Metabolism and nutrition disorders) | 48 (103)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 92 (452)
Blood uric acid increased (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 8 (10)
Iron overload (Metabolism and nutrition disorders) | 1 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 56 (167)
Serum calcium decreased (Metabolism and nutrition disorders) | 69 (236)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (15)
Serum glucose decreased (Metabolism and nutrition disorders) | 16 (31)
Serum magnesium decreased (Metabolism and nutrition disorders) | 43 (80)
Serum magnesium increased (Metabolism and nutrition disorders) | 24 (29)
Serum phosphate decreased (Metabolism and nutrition disorders) | 40 (102)
Serum potassium decreased (Metabolism and nutrition disorders) | 77 (270)
Serum potassium increased (Metabolism and nutrition disorders) | 16 (20)
Serum sodium decreased (Metabolism and nutrition disorders) | 43 (132)
Serum sodium increased (Metabolism and nutrition disorders) | 13 (20)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 17 (28)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (44)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arachnoiditis (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 5 (7)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 24 (39)
Dysgeusia (Nervous system disorders) | 8 (9)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 56 (113)
Intracranial hemorrhage (Nervous system disorders) | 2 (3)
Memory impairment (Nervous system disorders) | 2 (3)
Neuralgia (Nervous system disorders) | 6 (14)
Neurological disorder NOS (Nervous system disorders) | 8 (9)
Neuropathy - cranial (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 23 (57)
Peripheral sensory neuropathy (Nervous system disorders) | 50 (206)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1)
Sense of smell (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 6 (10)
Anxiety (Psychiatric disorders) | 21 (43)
Confusion (Psychiatric disorders) | 12 (13)
Depression (Psychiatric disorders) | 29 (56)
Insomnia (Psychiatric disorders) | 30 (50)
Libido decreased (Psychiatric disorders) | 2 (2)
Personality change (Psychiatric disorders) | 2 (3)
Psychosis (Psychiatric disorders) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 4 (7)
Dysuria (painful urination) (Renal and urinary disorders) | 7 (8)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 6 (7)
Incontinence (Renal and urinary disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (8)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 7 (12)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 4 (4)
Urogenital disorder (Renal and urinary disorders) | 9 (12)
Erectile dysfunction (Reproductive system and breast disorders) | 4 (4)
Gynecomastia (Reproductive system and breast disorders) | 2 (4)
Irregular menstruation (Reproductive system and breast disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 5 (5)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 2 (6)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (6)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 15 (33)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (75)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 22 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 (34)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 17 (23)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (56)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 13 (21)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (23)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 49 (78)
Skin disorder (Skin and subcutaneous tissue disorders) | 10 (12)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 32 (52)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (6)
Hemorrhage (Vascular disorders) | 8 (8)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 4 (4)
Hot flashes (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 27 (53)
Hypotension (Vascular disorders) | 23 (35)
Lymphedema (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (2)
Thrombosis (Vascular disorders) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval